CLINICAL TRIAL: NCT03515837
Title: A Randomized, Double-Blind, Phase 3 Study of Pemetrexed + Platinum Chemotherapy With or Without Pembrolizumab (MK-3475) in TKI-resistant EGFR-mutated Tumors in Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC) Participants (KEYNOTE-789)
Brief Title: Study of Pemetrexed + Platinum Chemotherapy With or Without Pembrolizumab (MK-3475) in Adults With Tyrosine Kinase Inhibitor- (TKI)-Resistant Epidermal Growth Factor Receptor- (EGFR)-Mutated Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC) (MK-3475-789/KEYNOTE-789)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-789; MK-3475-789 (Other: MSD); 184019 (Registry Identifier: JAPIC); 2017-004188-11 (EudraCT Number)
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Carboplatin; Cisplatin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembro+Pemetrexed+Chemo (Experimental): Participants receive pembrolizumab (pembro) 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W with no restrictions on the number of cycles PLUS platinum chemotherapy (chemo) (either carboplatin Area Under the Curve [AUC] 5 via IV infusion Q3W for 4 cycles [Cycles 1-4] or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles [Cycles 1-4]).
  Interventions: Biological: pembrolizumab; Drug: pemetrexed; Drug: carboplatin; Drug: cisplatin
- Placebo+Pemetrexed+Chemo (Active Comparator): Participants receive normal saline solution via IV infusion on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W with no restrictions on the number of cycles PLUS platinum chemotherapy (chemo)(either carboplatin AUC 5 via IV infusion Q3W for 4 cycles [Cycles 1-4] or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles [Cycles 1-4]).
  Interventions: Drug: pemetrexed; Drug: carboplatin; Drug: cisplatin; Drug: saline solution

INTERVENTIONS:
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475
  Arms: Pembro+Pemetrexed+Chemo
Drug: pemetrexed — IV infusion
Drug: carboplatin — IV infusion
Drug: cisplatin — IV infusion
Drug: saline solution — IV infusion
  Other Names: Normal saline solution
  Arms: Placebo+Pemetrexed+Chemo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pemetrexed plus platinum chemotherapy (carboplatin or cisplatin) with or without pembrolizumab (MK-3475; KEYTRUDA®) in the treatment of adults with the following types of tyrosine kinase inhibitor (TKI)-resistant, epidermal growth factor receptor (EGFR)-mutated, metastatic non-squamous non-small cell lung cancer (NSCLC) tumors: 1) TKI-failures (including osimertinib [TAGRISSO®] failure) with T790M-negative mutation tumors, 2) T790M-positive mutation tumors with prior exposure to osimertinib, and 3) first-line osimertinib failure regardless of T790M mutation status.

The primary study hypotheses are that the combination of pembrolizumab plus chemotherapy has superior efficacy compared to saline placebo plus chemotherapy in terms of: 1) Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) based on blinded independent central review, and 2) Overall Survival (OS). This study will be considered to have met its success criteria if the combination of pembrolizumab plus chemotherapy is superior to saline placebo plus chemotherapy in terms of PFS or OS.

Upon study completion, participants are discontinued and may be enrolled in a pembrolizumab extension study, if available.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of Stage IV non-squamous NSCLC.
* Documentation of tumor activating EGFR mutation, specifically either DEL19 or L858R.
* Investigator-determined radiographic disease progression per RECIST 1.1 after treatment with an EGFR TKI therapy: a) Participants previously treated with 1st or 2nd generation EGFR TKI (e.g. erlotinib/afatinib/gefitinib) are required to have confirmed documented absence of EGFR T790M mutation; b) Participants with confirmed acquired T790M mutation after 1st or 2nd generation EGFR TKI (e.g. erlotinib/afatinib/gefitinib) are required to have osimertinib TKI treatment failure prior to enrollment; c) Participants previously failed osimertinib TKI treatment as 1st line therapy are eligible regardless of their EGFR T790M mutation status. Note: TKI washout period for all participants is 1 week or 2 half-lives after last treatment dose, whichever is longer. TKI washout should be completed prior to first dose of study treatment.
* Measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology.
* Provided archival tumor tissue sample or newly obtained (no anti-neoplastic therapy since biopsy) core or excisional biopsy of a tumor lesion not previously irradiated.
* Life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to the first dose of study treatment but before randomization.
* Male participants must agree to use contraception during the treatment period and for at least 120 days after the last dose of pembrolizumab and up to 180 days after last dose of chemotherapeutic agents.
* Female participants must not be pregnant, not breastfeeding, and must agree to use contraception during the treatment period and for at least 120 days after the last dose of pembrolizumab and up to 180 days after the last dose of chemotherapeutic agents.
* Adequate organ function.

Exclusion Criteria:

* Predominantly squamous cell histology NSCLC. Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the participant is ineligible.
* Symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
* Received prior therapy with an anti-programmed cell death protein-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein-4 [CTLA-4], OX-40, CD137).
* Received prior systemic cytotoxic chemotherapy or investigational agent(s), excluding EGFR TKIs, for metastatic NSCLC. [Notes: 1) Prior treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic NSCLC. 2) If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment. 3) Prior exposure to traditional medicine(s) is allowed as long as therapy was discontinued at least 4 weeks prior to the first dose of study treatment.]
* Received prior radiotherapy within 2 weeks of start of study treatment or has received lung radiation therapy of >30 Gray (Gy) within 6 months before the first dose of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* Received a live vaccine within 30 days prior to the first dose of study treatment.
* Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment.
* Known additional malignancy that is progressing or has required active treatment within the past 5 years. (Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.)
* Known active untreated CNS metastases and/or carcinomatous meningitis.
* Severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* Known sensitivity to any component of cisplatin, carboplatin, or pemetrexed.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Active infection requiring systemic therapy.
* Known history of human immunodeficiency virus (HIV) infection.
* Known history of Hepatitis B or known active Hepatitis C virus.
* Known history of active tuberculosis (TB; Bacillus tuberculosis)
* Pregnant, breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of pembrolizumab and up to 180 days after the last dose of chemotherapeutic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (158):
- United States (19):
  - Cedars-Sinai Medical Center ( Site 0070), Los Angeles, California
  - Pacific Cancer Care ( Site 0058), Monterey, California
  - UC Irvine Medical Center/Chao Family Comprehensive Cancer Center ( Site 0092), Orange, California
  - St. Joseph Heritage Healthcare ( Site 0003), Santa Rosa, California
  - North Shore University Health System ( Site 0030), Evanston, Illinois
  - Siouxland Regioinal Cancer Center dba June E. Nylen Cancer Center ( Site 0065), Sioux City, Iowa
  - Southdale Cancer Care, University of Minnesota Medical Center- Edina ( Site 0048), Edina, Minnesota
  - Saint Lukes Hospital of Kansas City ( Site 0060), Kansas City, Missouri
  - New York Oncology Hematology P.C ( Site 8000), Albany, New York
  - Monter Cancer Center ( Site 0054), Lake Success, New York
  - Memorial Sloan Kettering Cancer Center-Rockerfeller Patient Pavilion ( Site 0049), New York, New York
  - White Plains Hospital Center for Cancer Care ( Site 0014), White Plains, New York
  - Providence Portland Medical Center ( Site 0097), Portland, Oregon
  - Kaiser Permanente Northwest ( Site 0037), Portland, Oregon
  - Parkland Health & Hospital System ( Site 2102), Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas ( Site 0035), Dallas, Texas
  - Utah Cancer Specialists ( Site 0001), Salt Lake City, Utah
  - Emily Couric Clinical Cancer Center ( Site 0020), Charlottesville, Virginia
  - Froedtert Hospital & the Medical College of Wisconsin ( Site 0041), Milwaukee, Wisconsin
- Australia (4):
  - Chris OBrien Lifehouse ( Site 0200), Camperdown, New South Wales
  - Westmead Hospital ( Site 0201), Westmead, New South Wales
  - Eastern Health ( Site 0202), Box Hill, Victoria
  - Austin Health ( Site 0203), Heidelberg, Victoria
- Brazil (8):
  - Liga Norte Riograndense Contra o Cancer ( Site 1909), Natal, Rio Grande do Norte
  - Hospital de Caridade de Ijui ( Site 1907), Ijuí, Rio Grande do Sul
  - Hospital Bruno Born ( Site 1913), Lajeado, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre ( Site 1905), Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 1904), Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos ( Site 1911), Barretos, São Paulo
  - Hosp. Clinicas da Fac. de Medicina de Ribeirao Preto - USP ( Site 1912), Ribeirão Preto, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 1903), São Paulo
- Canada (4):
  - William Osler Health System ( Site 0100), Brampton, Ontario
  - Sunnybrook Health Sciences, Odette Cancer Centre ( Site 0102), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0104), Toronto, Ontario
  - Jewish General Hospital ( Site 0105), Montreal, Quebec
- China (21):
  - The First Affiliated Hospital of Anhui Medical University ( Site 0721), Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 0717), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 0703), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0718), Beijing, Beijing Municipality
  - Southwest Hospital, The Third Military Medical University ( Site 0725), Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital ( Site 0723), Fuzhou, Fujian
  - The Affiliated Tumour Hospital of Harbin Medical University ( Site 0706), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0711), Zhengzhou, Henan
  - Xiangya Hospital of Central South University ( Site 0710), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0722), Changsha, Hunan
  - Jiangsu Cancer Hospital ( Site 0719), Nanjing, Jiangsu
  - The First Hospital of Jilin University ( Site 0702), Changchun, Jilin
  - Jilin Cancer Hospital ( Site 0705), Changchun, Jilin
  - Shanghai Chest Hospital ( Site 0700), Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University ( Site 0712), Shanghai, Shanghai Municipality
  - Tangdu Hospital ( Site 0708), Xi’an, Shanxi
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0709), Xi’an, Shanxi
  - Affiliated Tumor Hospital of Xinjiang Medical University ( Site 0701), Ürümqi, Xinjiang
  - The First Affiliated Hospital.Zhejiang University ( Site 0713), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital School of Medicine, Zhejiang University ( Site 0715), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0716), Hangzhou, Zhejiang
- France (9):
  - Centre Leon Berard ( Site 0801), Lyon, Auvergne
  - CHU Caen Service de Pneumologie ( Site 0804), Caen, Calvados
  - Centre Georges Francois Leclerc ( Site 0809), Dijon, Cote-d'Or
  - Hopital Jean Minjoz Besancon ( Site 0805), Besançon, Doubs
  - Hopital Prive d'Antony ( Site 0811), Antony, Hauts-de-Seine
  - C.H.U. de Tours - Hopital Bretonneau ( Site 0806), Tours, Indre-et-Loire
  - Centre D Oncologie de Gentilly ( Site 0810), Nancy, Meurthe-et-Moselle
  - Clinique Victor Hugo ( Site 0802), Le Mans, Sarthe
  - CHU Poitiers ( Site 0803), Poitiers, Vienne
- Germany (9):
  - Robert Bosch Krankenhaus Klinik Schillerhoehe ( Site 0904), Gerlingen, Baden-Wurttemberg
  - Universitaetsklinikum Mannheim ( Site 0911), Mannheim, Baden-Wurttemberg
  - Klinikum Wuerzburg Mitte gGmbH ( Site 0901), Würzburg, Bavaria
  - Pius Hospital Oldenburg ( Site 0905), Oldenburg, Lower Saxony
  - Florence Nightingale Krankenhaus ( Site 0912), Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte ( Site 0900), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Muenster ( Site 0906), Münster, North Rhine-Westphalia
  - Medizinische Fakultaet Carl Gustav Carus der TU Dresden ( Site 0907), Dresden, Saxony
  - Asklepios Klinikum Hamburg ( Site 0908), Hamburg
- Hong Kong (5):
  - Hong Kong Integrated Oncology Centre ( Site 0304), Hong Kong
  - Queen Mary Hospital ( Site 0301), Hong Kong
  - Queen Mary Hospital ( Site 0303), Hong Kong
  - Hong Kong United Oncology Centre ( Site 0306), Kowloon
  - Tuen Mun Hospital ( Site 0305), Tuenmen
- Israel (8):
  - Meir Medical Center ( Site 1701), Kfar Saba, Central District
  - Rabin Medical Center ( Site 1704), Petah Tikva, Central District
  - Rambam Medical Center ( Site 1703), Haifa, Heifa
  - Ha Emek Medical Center ( Site 1707), Afula, Northern District
  - Barzilai Medical Center ( Site 1706), Ashkelon, Southern District
  - Soroka Medical Center ( Site 1702), Beersheba, Southern District
  - Chaim Sheba Medical Center. ( Site 1700), Ramat Gan, Tell Abib
  - Sourasky Medical Center ( Site 1705), Tel Aviv, Tell Abib
- Italy (7):
  - Istituto Europeo di Oncologia ( Site 1303), Milan, Lombardy
  - Ospedale San Vincenzo di Taormina ( Site 1302), Taormina, Messina
  - AOU San Luigi Gonzaga di Orbassano ( Site 1300), Orbassano, Torino
  - IRCCS Giovanni Paolo II. Ospedale Oncologico ( Site 1305), Bari
  - Azienda Ospedaliero Universitaria Careggi ( Site 1301), Florence
  - Azienda Ospedaliera dei Colli V. Monaldi ( Site 1306), Napoli
  - Universita Campus Bio-Medico di Roma ( Site 1304), Roma
- Japan (19):
  - National Hospital Organization Nagoya Medical Center ( Site 0608), Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital ( Site 0612), Nagoya, Aichi-ken
  - Fujita Health University Hospital ( Site 0619), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 0601), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0616), Matsuyama, Ehime
  - Hyogo Cancer Center ( Site 0604), Akashi, Hyōgo
  - Kanazawa University Hospital ( Site 0617), Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center ( Site 0609), Yokohama, Kanagawa
  - Kansai Medical University Hospital ( Site 0606), Hirakata, Osaka
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0602), Sunto-gun, Shizuoka
  - National Hospital Organization Kyushu Medical Center ( Site 0621), Fukuoka
  - Kyushu University Hospital ( Site 0605), Fukuoka
  - Niigata Cancer Center Hospital ( Site 0610), Niigata
  - Okayama University Hospital ( Site 0614), Okayama
  - Osaka International Cancer Institute ( Site 0611), Osaka
  - National Cancer Center Hospital ( Site 0603), Tokyo
  - Toranomon Hospital ( Site 0615), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 0618), Tokyo
  - Wakayama Medical University Hospital ( Site 0613), Wakayama
- Mexico (4):
  - Instituto Jaliscience de Cancerologia ( Site 2000), Guadalajara, Jalisco
  - Medica Sur S.A.B de C.V. ( Site 2003), Mexico City
  - Oaxaca Site Management Organization SC ( Site 2001), Oaxaca City
  - Instituto Nacional de Cancerologia. ( Site 2007), Tlalpan
- South Korea (9):
  - Chungbuk National University Hospital ( Site 0404), Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Gachon University Gil Medical Center ( Site 0408), Incheon, Incheon-gwangyeoksi [Incheon]
  - National Cancer Center ( Site 0400), Gyeonggi-do, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0405), Seongnam-si, Kyonggi-do
  - Seoul National University Hospital ( Site 0402), Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center ( Site 0407), Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center ( Site 0403), Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic University of Korea. Seoul St. Mary s Hospital ( Site 0406), Seoul, Seoul-teukbyeolsi [Seoul]
  - Ulsan University Hospital ( Site 0401), Ulsan, Ulsan-Kwangyokshi
- Spain (7):
  - Hospitalo Univ. Germans Trias i Pujol ( Site 1100), Badalona, Barcelona [Barcelona]
  - Hospital de la Santa Creu i Sant Pau ( Site 1102), Barcelona, Barcelona [Barcelona]
  - Hospital Universitari Vall d Hebron ( Site 1106), Barcelona, Barcelona [Barcelona]
  - Hospital Ramon y Cajal ( Site 1101), Madrid
  - Hospital Universitario 12 de Octubre ( Site 1103), Madrid
  - Complejo Hospitalario Carlos Haya de Malaga ( Site 1107), Málaga
  - Hospital Universitario Virgen Macarena ( Site 1104), Seville
- Sweden (4):
  - Linkopings Universitetssjukhus ( Site 1504), Linköping, Ostergotlands Lan [se-05]
  - Skanes Universitetssjukhus Lund ( Site 1503), Lund, Skane Lan [se-12]
  - Karolinska Universitetssjukhuset Solna ( Site 1500), Solna, Stockholms Lan [se-01]
  - Sahlgrenska Universitetssjukhuset ( Site 1502), Gothenburg, Vastra Gotalands Lan [se-14]
- Taiwan (13):
  - Hualien Tzu Chi Medical Center-Hospital ( Site 0510), Hualien City, Hualien
  - Taipei Tzu Chi Hospital ( Site 0512), New Taipei City, New Taipei
  - Changhua Christian Hospital ( Site 0509), Changhua
  - National Taiwan University Hospital Hsin-Chu Branch ( Site 0511), Hsinchu
  - Kaohsiung Chang Gung Memorial Hospital ( Site 0507), Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital ( Site 0508), New Taipei City
  - China Medical University Hospital ( Site 0505), Taichung
  - Taichung Veterans General Hospital ( Site 0504), Taichung
  - National Cheng Kung University Hospital ( Site 0506), Tainan
  - National Taiwan University Hospital ( Site 0500), Taipei
  - Mackay Memorial Hospital ( Site 0503), Taipei
  - Taipei Veterans General Hospital ( Site 0501), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0502), Taoyuan District
- United Kingdom (8):
  - Sussex University Hospitals ( Site 1003), Brighton, Brighton And Hove
  - Western General Hospital ( Site 1009), Edinburgh, Edinburgh, City of
  - Leicester Royal Infirmary ( Site 1000), Leicester, Leicestershire
  - University College London Hospitals NHS Foundation Trust ( Site 1006), London, London, City of
  - Chelsea & Westminster Hospital ( Site 1001), London, London, City of
  - Birmingham Heartlands Hospital ( Site 1002), Birmingham
  - St James s University Hospital ( Site 1008), Leeds
  - Barking Havering and Redbridge University Hospitals NHS Trust Queen s Hospital ( Site 1004), Romford

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Yang JC, Lee DH, Lee JS, Fan Y, de Marinis F, Iwama E, Inoue T, Rodriguez-Cid J, Zhang L, Yang CT, de la Mora Jimenez E, Zhou J, Perol M, Lee KH, Vicente D, Ichihara E, Riely GJ, Luo Y, Chirovsky D, Pietanza MC, Bhagwati N, Lu S. Phase III KEYNOTE-789 Study of Pemetrexed and Platinum With or Without Pembrolizumab for Tyrosine Kinase Inhibitor-Resistant, EGFR-Mutant, Metastatic Nonsquamous Non-Small Cell Lung Cancer. J Clin Oncol. 2024 Dec;42(34):4029-4039. doi: 10.1200/JCO.23.02747. Epub 2024 Aug 22. PMID 39173098
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26126&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembro + Pemetrexed + Chemo: Participants received pembrolizumab (pembro) 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W with no restrictions on the number of cycles PLUS platinum chemotherapy (chemo) (either carboplatin Area Under the Curve [AUC] 5 via IV infusion Q3W for 4 cycles [Cycles 1-4] or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles [Cycles 1-4]).
- Placebo + Pemetrexed + Chemo: Participants received normal saline solution via IV infusion on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W with no restrictions on the number of cycles PLUS platinum chemotherapy (chemo)(either carboplatin AUC 5 via IV infusion Q3W for 4 cycles [Cycles 1-4] or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles [Cycles 1-4]). Eligible participants who had BICR-verified progressive disease were eligible to switch over to pembrolizumab monotherapy 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles.
Period: Overall Study
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Started | 245 | 247
Treated | 245 | 246
Switched Over to Pembro Monotherapy | 0 | 50
Completed | 0 | 0
Not Completed | 245 | 247
Not completed — Death | 219 | 227
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Participation Was Terminated By Sponsor | 26 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo | Total
Number analyzed (Participants) | 245 | 247 | 492
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (10.9) | 63.1 (10.0) | 62.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 151 | 303
  Male | 93 | 96 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 35
  Not Hispanic or Latino | 222 | 221 | 443
  Unknown or Not Reported | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 165 | 163 | 328
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 67 | 72 | 139
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 7 | 4 | 11
Geographic Region [Number; unit: Count of Participants] — Participants were stratified by geographic area of the enrolling site: East Asia versus Non-East Asia
  Count of Participants
    East Asia | 150 | 150 | 300
    Non-East Asia | 95 | 97 | 192
    EU | 53 | 47 | 100
    Non-EU | 192 | 200 | 392
    US | 3 | 6 | 9
    Non-US | 242 | 241 | 483
Programmed Death Ligand 1 (PD-L1) Status [Number; unit: Count of Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. PD-L1 status is determined by tumor proportion score (TPS). Participants with a TPS ≥50% were classified as PD-L1 strongly positive and participants with a TPS <50% were classified as not strongly positive.
  Count of Participants
    TPS ≥ 50% | 52 | 51 | 103
    TPS <50% | 181 | 185 | 366
    TPS ≥1% AND ≤49% | 54 | 72 | 126
    TPS <1% | 127 | 113 | 240
    Not evaluable | 12 | 11 | 23
Previous use of Tyrosine Kinase Inhibitor (TKI) Treatment History with Osimertinib [Number; unit: Count of Participants] — Participants were stratified using previous treatment history with TKI osimertinib: osimertinib or no osimertinib.
  Count of Participants
    Treated with TKI except for Osimertinib | 128 | 126 | 254
    Treated with first line Osimertinib | 28 | 33 | 61
    Treated with second line Osimertinib | 88 | 88 | 176
    Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PFS was assessed by blinded independent central review (BICR) using RECIST 1.1. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions is also considered PD. The PFS presented was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to ~40 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Number analyzed (Participants) | 245 | 247
Months | 5.6 [5.5 to 5.8] | 5.5 [5.4 to 5.6]
Statistical Analysis 1: Comparison: Pembro + Pemetrexed + Chemo vs Placebo + Pemetrexed + Chemo; Test type: Superiority; p = 0.0122, Log Rank; One-sided p-value based on log-rank test stratified by PD-L1 expression; treatment history; geographic region of the enrolling site; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.65 to 0.97] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by PD-L1 expression; treatment history; geographic region of the enrolling site

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis will be censored at the date of the last follow-up. The OS presented was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to ~51 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Number analyzed (Participants) | 245 | 247
Months | 15.9 [13.7 to 18.8] | 14.7 [12.7 to 17.1]
Statistical Analysis 1: Comparison: Pembro + Pemetrexed + Chemo vs Placebo + Pemetrexed + Chemo; Test type: Superiority; p = 0.0362, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.02] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1
Description: ORR was assessed by BICR using RECIST 1.1. ORR is defined as the percentage of participants in the analysis population who experience a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The ORR for participants is presented.
Time Frame: Up to ~51 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Number analyzed (Participants) | 245 | 247
Percentage of Participants | 29.0 [23.4 to 35.1] | 27.1 [21.7 to 33.1]
Statistical Analysis 1: Comparison: Pembro + Pemetrexed + Chemo vs Placebo + Pemetrexed + Chemo; Test type: Superiority; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-6.0 to 9.9] — Based on Miettinen & Nurminen method stratified by PD-L1 expression; treatment history; geographic region of the enrolling site

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1
Description: DOR was assessed by BICR using RECIST 1.1. For participants who experience a response of CR or PR, DOR is defined as the time from the earliest date of qualifying response until earliest date of PD or death from any cause, whichever comes first. The DOR presented was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to ~51 months
Population: All randomized participants that had a response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Number analyzed (Participants) | 245 | 246
Months | 6.3 [5.9 to 8.3] | 5.6 [4.4 to 6.3]

5. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are each scored on a 7-point scale (1=Very poor to 7=Excellent). The two raw scores were averaged into a combined score, then normalized using linear transformation so each participant's score ranged from 0 to 100 (0=Worst overall health/quality of life and 100=Best overall health/quality of life). The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score is presented.
Time Frame: Baseline and Week 18
Population: All randomized participants who had at least 1 patient reported outcome (PRO) assessment available and had received at least 1 dose of study intervention
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Number analyzed (Participants) | 241 | 243
Score on a Scale | -0.46 [-3.17 to 2.25] | -2.05 [-4.74 to 0.64]
Statistical Analysis 1: Comparison: Pembro + Pemetrexed + Chemo vs Placebo + Pemetrexed + Chemo; Test type: Other; Difference in LS Means = 1.59, 95% CI 2-sided [-1.93 to 5.10] — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by time interaction, stratification factors PD-L1 expression, treatment history, and geographic region of the enrolling site as covariates

6. Secondary Outcome: Time to True Deterioration (TTD) in the EORTC Questionnaire Composite Endpoint of Cough, Chest Pain or Dyspnea
Description: TTD is the time from baseline to first onset of 10 points or more deterioration from baseline with confirmation by the subsequent visit of 10 points or more deterioration from baseline in the composite endpoint of cough [EORTC QLQ-Lung Cancer Module 13 (LC13) Item 1; How much did you cough?], chest pain [EORTC QLQ-LC13 Item 10; Have you had pain in your chest?], or dyspnea [EORTC QLQ-C30 Item 8; Were you short of breath?]. Individual responses are given on a 4-point scale (1=Not at all; 4=Very much), with a lower score indicating a better outcome. The TTD was analyzed using the product-limit (Kaplan-Meier) method for censored data. The time to true deterioration in the composite endpoint of cough, chest pain or dyspnea is presented.
Time Frame: Baseline and up to ~51 months
Population: All randomized participants who had at least 1 PRO assessment available and had received at least 1 dose of study intervention
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Number analyzed (Participants) | 237 | 236
Months | NA [10.05 to NA] — NA = Median and upper range time to deterioration were not reached. | 17.97 [6.67 to NA] — NA = Upper range time to deterioration was not reached.
Statistical Analysis 1: Comparison: Pembro + Pemetrexed + Chemo vs Placebo + Pemetrexed + Chemo; Test type: Other; Hazard Ratio (HR) = 0.93, 95% CI [0.68 to 1.27] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of study treatment. The percentage of participants who experienced an AE is presented.
Time Frame: Up to ~44 months
Population: All randomized participants who received at least 1 dose of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Number analyzed (Participants) | 245 | 246
Percentage of Participants | 97.6 | 98.0

8. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to AEs
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of study treatment. The percentage of participants who discontinued study treatment due to an adverse event is presented.
Time Frame: Up to ~41 months
Population: All randomized participants who received at least 1 dose of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo
Number analyzed (Participants) | 245 | 246
Percentage of Participants | 19.2 | 17.1

ADVERSE EVENTS:
Time Frame: Death and Adverse Events up to ~59 months.
Description: Serious and Other adverse events (AEs) includes all participants who received ≥1 dose of study drug. All-Cause Mortality includes all randomized participants. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Groups:
- Placebo + Pemetrexed + Chemo Switched Over to Pembro Monotherapy: Participants who received placebo + pemetrexed + chemo per their randomized treatment assignment and had BICR-verified progressive disease were eligible to receive pembrolizumab monotherapy 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles.
Arm/Group | Pembro + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo | Placebo + Pemetrexed + Chemo Switched Over to Pembro Monotherapy
All-Cause Mortality (participants affected / at risk) | 219/245 | 186/247 | 44/50
Serious Adverse Events (participants affected / at risk) | 86/245 | 70/246 | 8/50
Other Adverse Events (participants affected / at risk) | 233/245 | 225/246 | 31/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Pemetrexed + Chemo (N=245) | Placebo + Pemetrexed + Chemo (N=246) | Placebo + Pemetrexed + Chemo Switched Over to Pembro Monotherapy (N=50)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 8 (8) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 3 (3) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 4 (6) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 5 (5) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 2 (3) | 0 (0)
Platelet count decreased (Investigations) | 8 (9) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 5 (5) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Pemetrexed + Chemo (N=245) | Placebo + Pemetrexed + Chemo (N=246) | Placebo + Pemetrexed + Chemo Switched Over to Pembro Monotherapy (N=50)
Anaemia (Blood and lymphatic system disorders) | 99 (161) | 110 (177) | 4 (4)
Hyperthyroidism (Endocrine disorders) | 13 (25) | 3 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 14 (18) | 6 (9) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 15 (15) | 2 (2)
Constipation (Gastrointestinal disorders) | 81 (124) | 76 (103) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 24 (27) | 18 (23) | 0 (0)
Nausea (Gastrointestinal disorders) | 96 (242) | 107 (237) | 4 (4)
Vomiting (Gastrointestinal disorders) | 48 (61) | 44 (55) | 5 (5)
Asthenia (General disorders) | 29 (41) | 28 (31) | 0 (0)
Chest pain (General disorders) | 17 (17) | 9 (10) | 3 (3)
Fatigue (General disorders) | 60 (81) | 49 (81) | 1 (1)
Malaise (General disorders) | 18 (31) | 23 (30) | 1 (1)
Oedema peripheral (General disorders) | 28 (42) | 24 (28) | 1 (2)
Pyrexia (General disorders) | 33 (54) | 21 (29) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 18 (21) | 2 (2)
Urinary tract infection (Infections and infestations) | 18 (19) | 13 (13) | 0 (0)
Alanine aminotransferase increased (Investigations) | 60 (96) | 58 (82) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 55 (98) | 55 (83) | 3 (3)
Blood creatinine increased (Investigations) | 24 (32) | 20 (23) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 19 (26) | 13 (14) | 4 (5)
Lymphocyte count decreased (Investigations) | 16 (20) | 11 (12) | 0 (0)
Neutrophil count decreased (Investigations) | 90 (236) | 113 (282) | 2 (2)
Platelet count decreased (Investigations) | 49 (81) | 52 (94) | 0 (0)
Weight decreased (Investigations) | 24 (29) | 16 (18) | 3 (3)
White blood cell count decreased (Investigations) | 71 (211) | 87 (259) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 64 (81) | 61 (79) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (16) | 18 (32) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (25) | 13 (19) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (20) | 21 (22) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (36) | 25 (29) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 17 (19) | 0 (0)
Dizziness (Nervous system disorders) | 22 (42) | 23 (38) | 1 (1)
Dysgeusia (Nervous system disorders) | 16 (35) | 6 (7) | 0 (0)
Headache (Nervous system disorders) | 29 (32) | 31 (33) | 0 (0)
Insomnia (Psychiatric disorders) | 23 (24) | 17 (17) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 41 (54) | 32 (36) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 21 (24) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (18) | 13 (15) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 12 (17) | 14 (16) | 3 (3)
Hypertension (Vascular disorders) | 11 (16) | 14 (15) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 (13) | 12 (14) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT03515837/Prot_SAP_001.pdf